CLINICAL TRIAL: NCT05623631
Title: Delphi Study to Identif Crucial Steps and Errors in the Placement of Chest Tubes
Brief Title: Delphi Study to Identify Crucial Steps and Errors in the Placement of Chest Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-09710
Record Dates: First submitted 2022-11-08; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Thoracic Injury
Keywords: Assessment; Chest Tube Insertion; Rating Scale
MeSH Terms: conditions — Thoracic Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delphi study (Other): Participants were asked to complete three rounds of surveys. These surveys collected information on which steps and errors can occur during CTI, and which of these should be included in an assessment tool.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Surveys were distributed using REDCap, and participants were asked to complete these within 5 weeks of receiving the invitation.

SUMMARY:
The goal of this Delphi study is to identify the crucial steps and the errors in Chest Tube Insertion (CTI). These steps and errors will be used for the development of a new assessment tool based on international consensus.

ELIGIBILITY:
Inclusion Criteria:

* Must be experts in their respective fields.
* Must hold a degree of Master in Medicine
* Must have finished the residency training specific to their field (be an attending physician)
* Must have 5 years post-residency experience
* Must have performed at least 50 CTIs independently in their career
* Must have an interest in educating and guiding junior residents in their training.

Exclusion Criteria:

* Insufficient experience in CTI
* Insufficient experience as an attending physician

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Steps and errors presented in round 1 | one year
  The number of experts who propose a certain step or error
Number of steps and errors passing round 2 | one year
  The number of experts who agree on the inclusion of each step or error in the assessment tool on a 5-point Likert scale (Strongly disagree - Disagree - Neutral - Agree - Strongly Agree).
Inclusion of steps with their descriptive anchors | one year
  The number of experts who agree on the inclusion of each step with their descriptive anchors in the assessment tool on a 5-point Likert scale (Strongly disagree - Disagree - Neutral - Agree - Strongly Agree).

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Willaert, Prof, Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium